CLINICAL TRIAL: NCT06420245
Title: A Prospective, Post-market Randomized Controlled Trial (RCT) to Demonstrate Clinical Utility of an Amniotic Membrane Allograft in Diabetic Foot Ulcer (DFU) Wound Management
Brief Title: Clinical Utility of an Amniotic Membrane Allograft for Diabetic Foot Ulcer Wound Management
Acronym: REBOUND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Medical Consultants (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LEGA-CLIN-2024-01
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: amniotic membrane allograft; diabetic foot ulcer; DFU
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Standard of care DFU wound management
  Interventions: Procedure: Standard of Care (SOC)
- Amniotic Membrane plus Standard of Care (Experimental): Weekly application of Orion™ amniotic membrane allograft in addition to standard of care DFU wound management
  Interventions: Device: Orion TM Amniotic Membrane Allograft; Procedure: Standard of Care (SOC)

INTERVENTIONS:
Device: Orion TM Amniotic Membrane Allograft — The intervention is a sterile allograft made from dehydrated extracellular matrix, designed to promote wound healing by providing a reliable and protective wound covering. Amniotic membranes are hypothesized to promote healing in open wounds by serving as a scaffold to support native tissue ingrowth, encouraging angiogenesis, and limiting microbial spread.
  Arms: Amniotic Membrane plus Standard of Care
Procedure: Standard of Care (SOC) — Standard wound care entails surgical debridement as needed to remove all non-viable tissue, screening for infection and probing of the wound for bone, weekly application of a collagen alginate primary dressing, and off-loading using a removable diabetic offloading cam-walker or total contact cast.

SUMMARY:
The goal of this clinical trial is to learn if use of Orion™, a dual-layer amniotic membrane allograft, in addition to standard wound care treatment can improve patient outcomes for people over the age of 50 with diabetic foot ulcers. The study aims to determine the incidence of complete wound closure at the end of 12 weeks of treatment. Researchers will compare the outcomes between a group of people treated with standard wound care and another group treated with standard wound care in addition to the amniotic membrane allograft to see if the amniotic membrane allograft improves wound healing.

During the study, participants will visit their doctor weekly over a 12 week period, which is standard for diabetic foot ulcer treatment procedures, and fill out a questionnaire measuring quality of life.

DETAILED DESCRIPTION:
Lower extremity diabetic ulcers are a common complication affecting millions of people in the United States. The purpose of this study is to evaluate the clinical utility of Orion™, a dual-layer amniotic membrane allograft, versus standard wound care in the management of diabetic foot ulcers. Amniotic membrane allografts are confirmed by the FDA Tissue Reference Group to meet the criteria for regulation solely under Section 361 of the PHS Act as defined in 21 CFR Part 1271 for the management of diabetic foot ulcers. Investigators hypothesize that the group of participants who receive amniotic membrane allografts in addition to standard wound care will experience a faster rate and higher incidence of complete wound closure compared to standard wound care alone. For only partially healed wounds, investigators anticipate a statistically significant reduction in the size of the ulcer and improved quality of life for participants in the experimental arm compared to standard wound care alone.

ELIGIBILITY:
Inclusion Criteria

1. Ambulatory patients ≥ 50 and ≤ 85 years of age;
2. Willing and able to provide informed consent;
3. Willing and able to comply with study requirements;
4. Presence of Wagner 1 and superficial Wagner 2 DFU extending at least through the dermis provided the DFU is located in the foot distal to the medial malleolus
5. If multiple Wagner 1 and superficial Wagner 2 DFUs are present, the largest ulcer meeting DFU eligibility criteria will be selected as the index DFU in the study;
6. Index ulcer is able to be visualized and accurately measured with eKare Insights;
7. Non-study ulcers must be > 2 cm (.79 in.) from the index ulcer;
8. Index DFU identified ≥ 4 weeks prior to study screening and < 52 weeks from the date of informed consent;
9. Index DFU area > 1.0 cm2 (0.39 in.) and < 25 cm2 (9.84 in.) at screening and at Wound Management Period Visit #1;
10. Index DFU offloaded according to SOC for entire run-in period, prior to randomization;
11. Potential participant is under the care of a clinician for diabetic management and other medical conditions (the site PI may assist/direct the patient in the pre-screening period to obtain a PCP).
12. Index foot has adequate circulation defined as meeting one (1) of the following within 30 days of screening:

A. ABI ≥ 0.7 and ≤ 1.3 AND TBI > 0.7; B. Dorsum transcutaneous oxygen tension measurement (TcPO2) ≥ 40 mmHg; C. Arterial duplex with biphasic flow in BOTH the DP and PT arteries verified by PI and documented.

Exclusion Criteria

1. Index foot ulcer documented to be caused by a medical condition other than diabetes;
2. Potential subject has five (5) or more DFUs and/or VLUs in the target limb;
3. DFU is secondary to Charcot neuroarthropathy;
4. Treatment with an antibiotic impregnated primary dressing ≤ 4 weeks prior to study screening;
5. Index ulcer is potentially or confirmed by biopsy to be cancerous;
6. Index ulcer site has undergone radiation therapy;
7. Venous leg ulcers in diabetic patients;
8. Active infection proximal to or at site of index ulcer;
9. Index foot ulcer reduced in area by ≥ 20% at the end of the 4-week run-in period;
10. Presence of active osteomyelitis or bone infection as verified by x-ray /MRI within 30 days of visit #1 of the run-in period;
11. Raynaud's disease;
12. Unreconstructible arterial ischemia which may lead to nonhealing;
13. Treatment with immunosuppressants, including systemic corticosteroids for ≥ 2 weeks within 30 days prior to study screening, or are anticipated during study participation;
14. Any active cancer undergoing treatment ≤ 30 days prior to wound management visit #1 of the run-in period, or is anticipated during study participation;
15. Treatment with chemotherapy within 30 days of the first study wound management visit of the run-in period, or is anticipated during study participation;
16. Diabetics with poor metabolic control, defined as HbA1c ≥ 12.0%, within 30 days of visit #1 of the run-in period;
17. Participation in an investigational device, biologic, or drug study currently or within 30 days of study wound management visit #1 of the run-in period;
18. Prior use of any advanced skin substitute product on the index ulcer within 60 days of visit #1 of the run-in period;
19. Index ulcer was continued to be treated after visit #1 of the run-in period and/or anticipate treatment during study participation with any of the following prohibited therapies:

    1. Biomedical or topical growth factor;
    2. Topical steroids applied to the index ulcer surface;
    3. On medications that are considered immune system modulators that could affect graft incorporation;
    4. Scarlet red dressing;
    5. Dakin's solution;
    6. Mafenide acetate;
    7. Tincoban;
    8. Zinc sulfate;
    9. Povidone-iodine solution;
    10. Polymyxin/nystatin;
    11. Chlorhexidine;
20. Patient is taking a cyclooxygenase-2 inhibitor (COX-2 inhibitor); such as, celecoxib (Celebrex, Consensi, Elyxyb), valdecoxib (Bextra), amlodipine (Consensi);
21. Patient has serum creatinine > 2.5 mg/dL within 30 days of study wound management visit #1 of the run-in period;
22. Autoimmune connective tissue disease;
23. End stage renal disease (ESRD);
24. Presence of any condition which would seriously compromise the subject's ability to complete this study;
25. Known history of poor adherence to medical therapy and/or clinic appointments;
26. Pregnant, or planning to become pregnant during the study;
27. Life expectancy < 1 year.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Complete Wound Closure | starting from randomization until last visit of the 12-week wound management period
  Percentage of enrolled study participants demonstrating 100% re-epithelialization of the index wound without leaking exudate at 12 weeks post-randomization.

SECONDARY OUTCOMES:
Time to complete wound closure | From time of randomization until the end of the twelve (12) week Wound Management Period.
  time to 100% re-epithelialization of the index ulcer without leaking exudate as assessed by Kare inSight®, starting at randomization through identification of complete wound closure.
Incidence of complete wound closure | From time of randomization to eight (8) weeks post-randomization.
  Incidence of complete wound closure, defined as 100% re-epithelialization of the index ulcer without leaking exudate as assessed by eKare inSight® at eight (8) weeks post-randomization.
Number of Orion™ Allografts or collagen alginate (SOC) dressings required for complete wound closure. | From the time of randomization through the twelve (12) week Wound Management Period.
  The number of Number of Orion™ Allografts or collagen alginate (SOC) dressings required for complete wound closure during twelve (12) week Wound Management Period.
Change in Quality of Life metrics | starting from randomization to last visit of the 12-week wound management period
  Change in QoL metrics at twelve (12) weeks post-randomization compared to baseline as reported by the subject in the WOUND-Q QoL questionnaires: Life Impact (8-32; higher is better); Lower Limb Symptoms (10-40; higher is better)
Recurrence Within Six Months | starting from last visit of the 12-week wound management period until 6-month follow-up visit
  Recurrence within six (6) months post wound managment period completion, defined as meeting the primary endpoint and reopening of index ulcer at the same site within six (6) months.
Change in wound size | from the time of randomization through twelve (12) weeks post-randomization.
  Percent area change of index ulcer at completion of twelve (12) weeks post-randomization.
Change in QoL metrics in follow-up. | From time of completion of the Wound Management Period through six (6) months.
  Change in QoL metrics to six (6) months after completion of the Wound Management Period as reported by the patient in the WOUND-Q QoL questionnaire.
Adverse events | From the time of randomization through six (6) month follow-up.
  Adverse events from randomization through six (6) month follow-up.
Serious adverse events | From the time of randomization through six (6) month follow-up.
  Occurrence of serious adverse events (SAEs) from randomization through six (6) month follow-up.
Major amputations | From the time of randomization through six (6) month follow-up.
  Major amputations defined as amputation above the metatarsals.
Minor amputations | From the time of randomization through six (6) month follow-up.
  Minor amputations defined as amputation involving toe or metatarsal only.
Hospital admission(s) | From the time of randomization through six (6) month follow-up.
  Hospital admission(s) and diagnosis from randomization through six (6) month follow-up.
Emergency Department (ED) visit(s) | From the time of randomization through six (6) month follow-up.
  ED visit(s) without admission through six (6) month follow-up.

OTHER OUTCOMES:
Per-Patient Product Cost | starting from randomization until last visit of the 12-week wound management period.
  Per-patient product cost for Orion™ Allografts during the course of wound management.
Number of wound management products used. | Following completion of the 12-week Wound Management Period (WMP Visit #13) through the six (6) month follow-up.
  Number of wound management products used in each group.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Clinical Research Inc., San Francisco, California
  - ILD Research Center, Vista, California

IPD SHARING:
Plan to Share IPD: Undecided